CLINICAL TRIAL: NCT04381078
Title: Does an Audio-visual Aid Reduce Anxiety and Improve the Understanding of Children Undergoing an Alveolar Bone Graft: Randomised Control Trial
Brief Title: Methods of Providing Information Prior to an Alveolar Bone Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18BA44
Record Dates: First submitted 2020-04-14; First posted 2020-05-08 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Cleft Lip and Palate
Keywords: cleft lip and palate; audiovisual guides; alveolar bone graft; anxiety
MeSH Terms: conditions — Cleft Lip; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Standardised Verbal Instructions Standardised Written Instructions Audiovisual Guide
  Interventions: Other: ACE - AudioVisual Guide
- Control (No Intervention): Standardised Verbal Instructions Standardised Written Instructions

INTERVENTIONS:
Other: ACE - AudioVisual Guide — Audiovisual guide to Alveolar Bone Graft Procedure, Pre-surgical orthodontics and post-operative care
  Arms: Intervention

SUMMARY:
Patients born with a cleft of the lip and/or palate may have a gap in the bone in the roof of their mouth and in the area of bone where the teeth develop. These patients require an alveolar bone graft (ABG) to allow the eruption of the maxillary canine teeth amongst other reasons. The optimal time to carry this out is between the ages of nine and eleven.

Whilst the patients will have had interventions as infants, this is often the first procedure a child born with a cleft lip and/or palate is likely to comprehend.

An audio-visual guide has been developed by the Great Ormond Street Hospital Dental Department for children undergoing an ABG. It explains the reason for the procedure, what the process will involve and advice regarding postoperative care.

This study will try ascertain whether providing information to patients and parents in this manner reduces anxiety, improves understanding of why the procedure was undertaken and post-operative care.

Children between the ages of eight and twelve ready for this procedure at Great Ormond Street Hospital will be enrolled. They will be allocated into two groups during their assessment appointment. The control will be given standardised verbal and written information, whilst the experimental group will also be given the animation. The level of anxiety and understanding of the procedure will be measured after the intervention/control information and once again when the patient attends for their pre-surgical assessment two to three months later.

This study aims to see whether the patient and parent anxiety is reduced and knowledge regarding the procedure is improved when utilising this of kind audio-visual guide for children. This will indicate whether it is worthwhile committing resources to the development of similar animations for other procedures.

DETAILED DESCRIPTION:
Study Overview This is a single-centre prospective randomised control trial at (Great Ormond Street Hospital) with concealed allocation. A randomised controlled trial was chosen to allow equal distribution of confounding factors including age, gender and previous experience of orthodontic or surgical procedures.

Enrollment Patients identified by the cleft team as needing an alveolar bone graft are booked onto joint maxillofacial - orthodontic clinics which run several times a week. The clinical notes of these clinics will be screened for patients by a member of the study team (who are also part of the clinical care team) two weeks before a clinic The parents/guardian of patients identified as meeting the inclusion/exclusion criteria will be called by identified members of the research team to explain the study. They will seek consent for Patient Information Sheets (PIS) to be posted to their registered address at least one week before the appointment date (Appendix D&E).

On the day of the assessment, children deemed suitable will be invited to participate. The researcher will go through the PIS verbally in detail allowing the participants to ask any questions. Verbal and then written consent will be obtained from those willing to participate. They will be allocated into a control or intervention group using a random number generator to ensure a randomised and concealed allocation process.

The sample size calculation has been carried out, using previous studies that have used the primary outcome measure. 56 children will be recruited accounting for a 20% drop out rate.

The Null Hypothesis:

The "ACE" animation does not reduce the anxiety of patients between the age of eight and twelve years undergoing an alveolar bone graft (ABG).

Alternative Hypothesis:

The "ACE" animation reduces the anxiety of patients between the age of eight and twelve years undergoing an alveolar bone graft (ABG).

Intervention A control group will receive standardised verbal and written information (the current protocol). The study group will additionally be given the "ACE" animation.

A control arm will be utilised, so the investigators can ascertain if the animation does make a difference to the anxiety and understanding of children/adults. As the animation is not routinely provided to children, this group will not be disadvantaged when compared to our current practice and patient cohort.

However, if the alternative hypothesis is true the control group will be disadvantaged. The investigators will mitigate this by showing all those in the control group the animation (during the pre-assessment appointment).

Outcome Measures The primary outcome measure is the State Anxiety Section of State-Trait Anxiety Inventory for Children (STAIC -S)- a validated measure of child anxiety (Appendix B). This will be given to both groups on enrolment (T1) as a baseline. At the end of the assessment appointment during which participants will have received the control or intervention they will be asked to fill this questionnaire again (T2). The patient will be asked to fill this anxiety assessment when they attend for their pre-surgical assessment which is usually 2-3months later (T3). This will allow us to ascertain whether there is a short and/or long-term change in anxiety.

The secondary outcome measures will be assessed by the State Anxiety section of State-Trait Anxiety Inventory (Appendix Bii), to be filled in by the parents at the same time points (T1,T2,T3).

In addition, participants and parents of both intervention and control will fill in their respective parts of a questionnaire that assesses their self-reported understanding of the procedure (Appendix Ci and Cii). This will happen at time points T2 (end of assessment appointment) and T3(end of pre-surgical appointment).

This questionnaire has been developed by an expert panel of Consultant Orthodontists, Restorative Dentists, Paediatric dentists, Maxillofacial and Oral Surgeons and Clinical Psychologists, followed by a Patient and Public Involvement session with the GOSH London Young Person's Advisory Group - a group of 8 to 21 year olds.

This group was invited to recommend changes to the Participant Information Sheets, Consent/Assent forms and Questionnaires to improve their acceptability and readability. They were also asked to make changes to the questionnaire to better reflect what they wanted to know as patients and the public. Changes to the layout and wording were presented to the Expert panel and broadly accepted. The YPAG voted this project as being the most interesting and informative of their session.

Bias in the study will be minimised by randomisation and concealed allocation processes. Patients/parents will be blinded, they will not be told if they are in the control or intervention group. The Participant Information Sheets do not mention an animation.

Statistical analysis This will be undertaken by a statistician independent from the clinical care team who is blinded to which group is the intervention and the control.

A narrative description of the protocol is given in Appendix N.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of eight and twelve
* With Cleft lip and/or palate requiring and ready for an alveolar bone graft
* That consent to inclusion in the study
* Irrespective of gender.

Exclusion Criteria:

* Diagnosed Syndrome
* Identified global developmental delay
* Previous alveolar bone graft
* Patient and/or parent/guardian unable to read/understand English
* Declined to participate

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Section of State-Trait Anxiety Inventory for Children | Change from baseline to immediately after intervention, an average of 30minutes
  Validated measure of Child State Anxiety
State Anxiety Section of State-Trait Anxiety Inventory for Children | Change from baseline to surgical pre-assessment appointment, an average of 3months
  Validated measure of Child State Anxiety

SECONDARY OUTCOMES:
State Anxiety section of State-Trait Anxiety Inventory | Change from baseline to immediately after intervention, an average of 30minutes
  Validated measure of Adult State Anxiety
State Anxiety section of State-Trait Anxiety Inventory | Change from baseline to surgical pre-assessment appointment, an average of 3months
  Validated measure of Adult State Anxiety
Patient Questionnaire | Change from baseline to immediately after intervention an average of 30minutes
  Self-reported understanding of procedure
Patient Questionnaire | Change from baseline to surgical pre-assessment appointment, an average of 3months
  Self-reported understanding of procedure
Parent/Legal Guardian Questionnaire | Change from baseline to immediately after intervention an average of 30minutes
  Self-reported understanding of procedure
Parent/Legal Guardian Questionnaire | Change from baseline to surgical pre-assessment appointment, an average of 3months
  Self-reported understanding of procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No